CLINICAL TRIAL: NCT02303548
Title: Pilot Study of Bicarbonate Injection for Improving Outcome in Patients With Out-of-hospital Cardiac Arrest, Double-blind Randomized Control Trial
Brief Title: Bicarbonate in Patients With Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Won Young Kim, Associate proffesor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BicarbonateinCPR001
Record Dates: First submitted 2014-11-23; First posted 2014-12-01 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrest; Metabolic Acidosis
Keywords: Sodium Bicarbonate
MeSH Terms: conditions — Heart Arrest; Acidosis | interventions — Sodium Bicarbonate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Sodium bicarbonate) (Experimental): Sodium bicarbonate 50cc (50mEq) intravenous injection over 2 min
  Interventions: Drug: Sodium bicarbonate
- 2 (Normal saline) (Placebo Comparator): Normal saline 50cc intravenous injection over 2 min
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Sodium bicarbonate — Administer Sodium bicarbonate 50 mEq IV over 2 minutes
  Other Names: Bivon
  Arms: 1 (Sodium bicarbonate)
Drug: Normal saline — Placebo
  Other Names: 0.9% sodium chloride
  Arms: 2 (Normal saline)

SUMMARY:
A pilot study to evaluate the effect of sodium bicarbonate administration on cardiopulmonary resuscitation results and outcomes in cardiac arrest patient with severe metabolic acidosis.

ELIGIBILITY:
Inclusion Criteria:

* adult cardiac arrest patient with arterial pH <7.1 or bicarbonate <10mmEq/L checked at 10 minutes of cardiopulmonary resuscitation

Exclusion Criteria:

* age <18 trauma patient Do Not Resuscitate state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

REFERENCES:
- [Derived] Ahn S, Kim YJ, Sohn CH, Seo DW, Lim KS, Donnino MW, Kim WY. Sodium bicarbonate on severe metabolic acidosis during prolonged cardiopulmonary resuscitation: a double-blind, randomized, placebo-controlled pilot study. J Thorac Dis. 2018 Apr;10(4):2295-2302. doi: 10.21037/jtd.2018.03.124. PMID 29850134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 (Sodium Bicarbonate) | 2 (Normal Saline)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 (Sodium Bicarbonate) | 2 (Normal Saline) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (16.4) | 64.1 (15.4) | 64.8 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 18 | 21 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 25 | 25 | 50
pH [Median (Inter-Quartile Range); unit: units on a scale] | 6.99 [6.92 to 7.12] | 6.90 [6.85 to 6.94] | 6.95 [6.87 to 7.04]
Shockable pre-hospital rhythm [Number; unit: participants] — Shockable pre-hospital rhythm: ventricular fibrillation or pulseless ventricular tachycardia rhythm detection before hospital admission
  participants | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Return of Spontaneous Circulation (ROSC)
Description: Percentage of Participants with Return of Spontaneous Circulation (ROSC)
Time Frame: checked during CPR, duration of ROSC >20 min
Measure: Number; unit: ROSC percents of each group
Arm/Group | 1 (Sodium Bicarbonate) | 2 (Normal Saline)
Number analyzed (Participants) | 25 | 25
ROSC percents of each group | 4 | 16

ADVERSE EVENTS:
Arm/Group | 1 (Sodium Bicarbonate) | 2 (Normal Saline)
All-Cause Mortality (participants affected / at risk) | 24/25 | 21/25
Serious Adverse Events (participants affected / at risk) | 25/25 | 24/25
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (Sodium Bicarbonate) (N=25) | 2 (Normal Saline) (N=25)
Severe hypoxic brain injury (Nervous system disorders) | 25 (25) | 24 (24) — Severe cerebral disabilities which occurred due to hypoxic brain injury such as conscious, but dependent on others for daily support because of impaired brain function, coma or vegetative state, or brain death within 28 days
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (Sodium Bicarbonate) (N=25) | 2 (Normal Saline) (N=25)
Severe hypoxic brain injury (<6 mo) (Nervous system disorders) | 25 (25) | 25 (25) — Severe cerebral disabilities which occurred due to hypoxic brain injury such as conscious, but dependent on others for daily support because of impaired brain function, coma or vegetative state, or brain death within 6 months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes